CLINICAL TRIAL: NCT04571970
Title: A Phase I/II Multicenter, Open-Label Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of RGX-121 in Children 5 Years of Age and Older With MPS II (Hunter Syndrome)
Brief Title: RGX-121 Gene Therapy in Children 5 Years of Age and Over With MPS II (Hunter Syndrome)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: REGENXBIO Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGX-121-1102
Record Dates: First submitted 2020-09-23; First posted 2020-10-01 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Mucopolysaccharidosis Type II (MPS II)
Keywords: MPS II; gene therapy; Hunter
MeSH Terms: conditions — Mucopolysaccharidosis II; Sudden Infant Death

STUDY DESIGN:
Intervention Model Description: Single-arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): 6.5 × 10^10 GC/g brain mass of RGX-121
  Interventions: Genetic: RGX-121

INTERVENTIONS:
Genetic: RGX-121 — Recombinant adeno-associated virus serotype 9 capsid containing human iduronate-2-sulfatase expression cassette

SUMMARY:
RGX-121 is a gene therapy which is designed to deliver a functional copy of the iduronate-2-sulfatase (IDS) gene to the central nervous system. This study is a phase I/II study to determine whether RGX-121 is safe, well tolerated, and potentially effective in children five years of age and over who have severe MPS II.

DETAILED DESCRIPTION:
MPS II is a rare X-linked recessive genetic disease caused by mutations in the iduronate-2-sulfatase (IDS) gene. Enzyme replacement therapy (ERT) with recombinant idursulfase (ELAPRASE®) is the only approved product for the treatment of Hunter syndrome; however, ERT as currently administered does not cross the blood brain barrier and is therefore unable to address the unmet need in MPS II patients with CNS (neurocognition and behavior) involvement. RGX-121 is designed to deliver a healthy gene to cells in the CNS and iduronate-2-sulfatase (I2S) may then be secreted by transduced cells which may cross-correct non-transduced cells by taking up the functional enzyme. This is a Phase I/II, multicenter, open-label, single arm study of RGX-121. Approximately 6 children (≥ 5 years to < 18 years of age) who have severe (neuronopathic) MPS II could be enrolled into a single dose cohort and will receive a single dose of RGX-121 administered by IC or ICV injection. Safety will be the primary focus for the initial 24 weeks after treatment (primary study period). Following completion of the primary study period, participants will continue to be assessed (safety and efficacy) for up to a total of 104 weeks following treatment with RGX-121.

ELIGIBILITY:
Inclusion Criteria:

Meets any of the following criteria:

1. Has a documented diagnosis of MPS II AND a neurocognitive testing score ≤ 1 ½ standard deviation (SD) from the test normative mean (BSID-III: 77 and MSEL Visual Reception: 35), OR
2. Has a documented diagnosis of MPS II AND has a decline of ≥ 1 standard deviation on serial neurocognitive testing administered between 3 to 36 months apart (BSID-III Cognitive or MSEL Visual Reception), OR
3. Has a relative clinically diagnosed with neuronopathic MPS II who has the same IDS mutation as the participant AND the participant in the opinion of a geneticist has inherited a neuronopathic form of MPS II, OR
4. Has documented mutation(s) in IDS that in the opinion of a geneticist is known to result in a neuronopathic phenotype AND in the opinion of a clinician has a neuronopathic form of MPS II

Exclusion Criteria:

1. Has contraindications for intracisternal injection, intracerebroventricular injection, or lumbar puncture
2. Has contraindications for immunosuppressive therapy
3. Has any neurocognitive deficit not attributable to MPS II or diagnosis of a neuropsychiatric condition
4. Has had prior treatment with an AAV-based gene therapy product
5. If receiving ELAPRASE® via intrathecal (IT) administration, must agree to discontinue IT idursulfase for the duration of the study
6. Has experienced a serious hypersensitivity reaction to intravenous (IV) ELAPRASE®
7. Is currently failing to respond to idursulfase (ELAPRASE®) IV due to neutralizing anti-idursulfase antibodies
8. Has received any investigational product within 30 days of Day 1 or 5 half-lives before signing of the ICF, whichever is longer
9. Has a platelet count <100,000 per microliter (µL), absolute neutrophil count <1.0 × 103/µL, or aminotransferase (ALT) or aspartate aminotransferase (AST) >3 × upper limit of normal (ULN) or total bilirubin >1.5 × ULN at screening unless the participant has a previously known history of Gilbert's syndrome

Ages: 5 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events and serious adverse events | 24 Weeks
  Number of participants with treatment-related adverse events and serious adverse events as assessed by CTCAE (Version 5.0)

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events and serious adverse events | 104 Weeks
  Number of participants with treatment-related adverse events and serious adverse events as assessed by CTCAE (Version 5.0)
Biomarkers | Baseline, Week 1, Week 2, Week 4, Week 12, Week 24, Week 38, Week 52, Week 64, Week 78, Week 104
  Change from baseline in Glycosaminoglycan levels (ng/mL)
Biomarkers | Baseline, Week 1, Week 2, Week 4, Week 12, Week 24, Week 38, Week 52, Week 64, Week 78, Week 104
  Change from baseline in iduronate-2-sulfatase activity
Change in neurodevelopmental parameters | Baseline, Week 52, Week 104
  Change from baseline in neurodevelopmental parameters of cognitive function as measured by the Bayley Scales of Infant and Toddler Development, 3rd Edition (BSID-III)
Change in neurodevelopmental parameters | Baseline, Week 52, Week 104
  Change from baseline in neurodevelopmental parameters of cognitive function as measured by the Mullen Scales of Early Learning (MSEL)
Change in neurodevelopmental parameters | Baseline, Week 24, Week 52, Week 78, Week 104
  Change from baseline in neurodevelopmental parameters as measured by the Vineland Adaptive Behavior Scales, 2nd Edition (VABS-II), Comprehensive Interview Form

CONTACTS AND LOCATIONS:
Locations (2):
- University of California San Francisco, Benioff Children's Hospital, Oakland, California, United States
- McGill University Heath Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No